CLINICAL TRIAL: NCT00798564
Title: Explorative Study "Exercise Induced Asthma and Airway Reactivity in Athletes"
Brief Title: Exercise Induced Asthma and Airway Reactivity in Athletes
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Principal Investigator, Leif Bjermer, Professor, MD, Skane University Hospital
Other Study IDs: 34797
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Function Tests
Keywords: Exercise; Mannitol
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall aim is to explore pathophysiological factors related to airway hyperresponsiveness to direct and indirect provocation stimuli in athletes with different sport activities, with special focus on epithelial reaction linked to CC16 and to eicosanoid related inflammatory response. The investigators also wish to compare indirect testing done as hyper osmotic challenge with Mannitol compared to a defined sport specific exercise challenge.

DETAILED DESCRIPTION:
By non-invasive tools the investigators wish to characterize type of airway reaction to various provocative stimuli in athletes doing two different sort activities, Tennis or swimming. As controls are being used sedentary age-matched controls from the same region, exposed to the same school environment. Thus we wish to:

* explore the prevalence of positive mannitol reactivity among swimmers and tennis player and how this relates to symptoms, disease history and to a sport specific exercise provocation test.
* compare the results from sport specific testing with a standardized eucapnic hyperventilation test (EHV)
* compare the overall reactivity to mannitol or EHV among swimmers and tennis players compared to aged matched controls.
* explore the role by CC16 in airway reactivity to different provocative stimuli and to see whether there is a difference between different sport activities, different test protocols and between athletes and controls.
* explore evidence of eicosanoid related inflammatory reaction in athletes and controls in relation to different provocative stimuli

The study population consists of 100 elite swimmers, 100 elite tennis players and 100 non-elite, eged matched controls. In the latter group, 30 are aged matched non-atopic non-asthmatic controls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 16-19 from Skåne.
* All should approve attendance in the study by signing an informed consent. Igf they are aged under 18, parents should also sign.
* Three groups are included
* Elite aspiring swimmers with an average training intensity of at least hours per week the last year.

Exclusion Criteria:

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 100 elite swimmers 100 elite tennis players 100 aged matched non-atletic subjects, 30 aged-matcked healthy non-atopic controls
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leif H Bjermer, MD, PhD, Principal Investigator — Lund University